CLINICAL TRIAL: NCT07384884
Title: Surgery and Laser Interstitial Thermal Therapy for Bilateral Glioblastomas
Acronym: SLITT-GBM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 359416
Record Dates: First submitted 2025-08-11; First posted 2026-02-03 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Brain Tumours; GBM
Keywords: brain tumour
MeSH Terms: conditions — Brain Neoplasms | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Surgical resection followed by LITT (Other): Combined unilateral open surgery for maximal tumour resection followed by contralateral LITT to the smaller component/residual.
  Interventions: Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines

INTERVENTIONS:
Procedure: surgery (any volume) and / or pharmaceuticals treatment initiated or planned or only dynamic observation, in accordance with current clinical guidelines — All patients will have combined unilateral open surgery for maximal tumour resection followed by contralateral LITT to the smaller component/residual.
  Other Names: laser interstitial thermal therapy

SUMMARY:
Butterfly glioblastomas (bGBM), defined as tumours crossing the midline to involve hemispheres bilaterally, have a dismal prognosis with a median survival of 3.3-6 months and only 9% of patients with bGBM survive 2-years. These figures put bGBM in the worst end of the spectrum of GBM prognosis, significantly inferior to the survival figures quoted in the literature with standard of care - 14.6 months - particularly when 5-aminolevulinic acid is used as surgical adjuvant - 17.47 months.

Despite the poor outcome of this disease, there is preliminary evidence suggesting that active oncology treatment can impact the survival of patients with this condition.With particular regards to surgical resection versus biopsy, there is a suggestion that resection improves overall survival at 6 months with no clear difference at 12 and 18 months of follow up.

Laser-induced thermal therapy (LITT) is a minimally invasive laser ablation technique used in a range of brain tumours, including glioblastomas, with similar overall survival to the ones reported for open surgery in patients with lesions not amenable to open resection. The minimally invasive nature of this technique, significantly reducing the collateral damage to the surrounding brain structures, suggests Its potential in the treatment of this bGBM [14] with significant implications as a deficit-sparing technique, particularly if associated with preoperative and intraoperative monitoring and mapping techniques.

The SLITT-GBM study will combine unilateral open surgery for maximal tumour resection with contralateral LITT to the smaller component/residual.

ELIGIBILITY:
Inclusion Criteria:

1. Presumptive diagnosis of bGBM as per preoperative MRI and MDT assessment
2. Presumed residual / smaller component of the bGBM has to be < 2.5cm
3. Performance Status 0-1
4. Able to consent for the study

Exclusion Criteria:

1. bGBM measuring >2.5 cm in both hemispheres.
2. Tumour progression between surgical debulking and LITT treatment
3. Severe complications after surgery (hydrocephalus, infection, heamatoma, stroke)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Neurocognitive Function | 12 months
  To assess post-operative neurocognitive function using the Montreal Cognitive Assessment

SECONDARY OUTCOMES:
Progression-free survival in years | 12 months
  To evaluate progression-free survival
Assessing Quality of Life | 12 months
  To assess quality of life using the EORTC QLQ-C30 assessment

CONTACTS AND LOCATIONS:
Locations (1):
- King's College NHS Foundation Trust, London, United Kingdom